CLINICAL TRIAL: NCT05042583
Title: Effect of Ultrasound-guided Left Stellate Ganglion Block on Rapid Recovery in Patients With Liver Lobectomy and Its Mechanism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhonghua Chen,MD (Other)
Collaborators: China (Zhejiang) Health technology RESEARCH and development and transformation platform (Unknown)
Responsible Party: Sponsor-Investigator, Zhonghua Chen,MD, associate chief physician, Shaoxing Hospital of Zhejiang University
Organization: Shaoxing Hospital of Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2021-09-04; First posted 2021-09-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Left Stellate Ganglion Block on Rapid Recovery; Possible Molecular Mechanism of Left Stellate Ganglion Block
Keywords: Guided by ultrasound; Stellate ganglion block; hepatectomy; ERAS

STUDY DESIGN:
Intervention Model Description: Sixty patients with liver lobectomy were selected and divided into two groups according to random number table method: experimental group and control group., with 30 cases in each group. All enrolled patients signed informed consent. Control group: The control group was injected with physiological saline 6ml for stellate ganglion block.Experimental group: The experimental group was injected with 0.5% ropivacaine 6ml for stellate ganglion block.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the experimenters nor the participants knew whether they were getting an experimental drug or a placebo. In this way, the description of the therapeutic effects and adverse reactions of the subjects, as well as the record of the various reactions of the experimenters, can be as objective as possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group was injected with 0.5% ropivacaine 6ml
  Interventions: Procedure: Stellate ganglion block
- Control group (Placebo Comparator): control group was injected with 6ml normal saline.
  Interventions: Procedure: Stellate ganglion block

INTERVENTIONS:
Procedure: Stellate ganglion block — The probe direction was 30-45 degrees from the sagittal plane of the neck. The anterior nodules of the transverse process of the sixth cervical vertebra were displayed. The important anatomical structures were distinguished, and the internal carotid artery and longus cervical muscle were observed. A 25G, 6cm puncture needle was used with the tip beveled downward, and the needle path and tip were shown under ultrasound. The tip reached the high-echo sieve structure between the carotid artery and longus cervical muscle, and the drug solution was injected after withdrawal without blood and gas . The experimental group was injected with 6ml 0.5% ropivacaine.

SUMMARY:
Lobe resection of complex process Traumatic big liver door block causes the body's nervous system very excited or inhibit the endocrine system, immune excessive activation of inflammatory cells, triggering and cause dysfunction of the immune inflammatory reaction, of patients with injury of tissues and organs and affect its repair, increase the risk of complications after liver resection, affected lobe resection in patients with postoperative rapid recovery. Stellate ganglion block has been widely used in the treatment of various systemic diseases due to its advantages of simple operation and obvious effect. SGB has broad application prospects and can promote postoperative recovery of patients undergoing major surgery, but its effect on the rapid recovery of patients undergoing liver lobectomy and its mechanism remain to be further explored.

DETAILED DESCRIPTION:
Stellate ganglion, also known as cervicothoracic sympathetic ganglion, is a fusion of the subcervical sympathetic ganglion emitted from C3-C7 and the first thoracic sympathetic ganglion, located in the lateral lateral of the transverse tubercle of the 7th cervical vertebra and the cervical protubertion of the first rib, and receives THE T1-T2 nerve SGB, which is mainly manifested in the central and peripheral nerves The central function is to maintain the stability of internal environment by regulating the activity of hypothalamus. The peripheral effect is mainly manifested by blocking the preganglionic and postganglionic fibers, which inhibits the muscle tension, cardiovascular movement and bronchoconstrictor glands in the distribution area to secrete pain conduction, so as to achieve the purpose of treating diseases such as heart, lung, head and neck. The study also found that SGB can regulate the endocrine system autonomic nervous system and immune system, and play an important role in maintaining the stability of the body's internal environment. SGB is considered a very important weapon for modern anesthesiologists. The clinical application of SGB is not only for the pain treatment of head, face, neck, shoulder and limb, but also for the treatment of arrhythmia, traumatic stress and the control of hypertension. SGB has been shown to be effective in treating ventricular arrhythmias, stopping ventricular tachycardia in patients with long QT syndrome, and ventricular fibrillation with recurrent acute myocardial infarction. SGB has a certain therapeutic effect on pulmonary hypertension by down-regulating sympathetic activity and improving endothelial dysfunction. SGB can regulate gastrointestinal dysfunction, promote gastrointestinal motility recovery, and has obvious curative effect on gastrointestinal diseases. Studies have confirmed that SGB can significantly decrease serum inflammatory cytokines IL-1B,IL-6 and TNF-α. Planetary ganglion block in patients with severe trauma showed significant downregulation of inflammatory factors IL-1B,IL-6 and TNF-α in patients with 6, 24 and 72 hours, suggesting that SGB has a regulatory role in the early inflammatory response of trauma and improves the prognosis of acute trauma. SGB can reduce the inflammatory response, improve gastrointestinal dysfunction and promote the recovery of gastrointestinal function after surgery by reducing stress response, inhibiting the synthesis of cytokines inflammatory mediators and nitric oxide synthase

ELIGIBILITY:
Inclusion Criteria:Sixty patients with elective lobectomy； heart function grade I or II；ASA grade I or II；aged 18-70 years.

-

Exclusion Criteria:Non-lobectomy patients； age <18 and > 70 years old；heart function grade ≥ III, ASA grade ≥ III; Hypersensitivity to local anesthesia；combined with immune disease or immunosuppression;severe mental illness unable to cooperate with SGB;abnormal neck anatomy；Stellate ganglion block failure；the patient refused to participate in the study.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | Within one week after surgery
  pulmonary infection, oxygenation injury, arrhythmia, bleeding, intestinal paralysis, incision infection, renal insufficiency, cognitive dysfunction, etc.
mortality rate | Within 30 days after surgery
  mortality rate
Plasma concentrations of IL-6,IL-10 and TNF-α | Within three days of the surgery
  Plasma concentrations of IL-6,IL-10 and TNF-α were measured before operation, 6 h after operation, 24 h after operation, and 72 h after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoxing People's Hospital, Shaoxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lao WL, Sang S, Huang LC, Yi SH, Guo MC, Dong HM, Zhou GZ, Chen ZH. Effect of ultrasound-guided stellate ganglion block on inflammatory cytokines and postoperative recovery after partial hepatectomy: a randomised clinical trial. BMC Anesthesiol. 2024 Jan 2;24(1):7. doi: 10.1186/s12871-023-02392-7. PMID 38166634